CLINICAL TRIAL: NCT01593774
Title: Phase 2 Study of Melatonin Adjunct to Olanzapine for Prevention of Olanzapine-associated Metabolic Side Effects.
Brief Title: Melatonin for Prevention of Metabolic Side Effects of Olanzapine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Guilan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad Jafar Modabbernia, Associate Professor of Psychiatry, Guilan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GUMS-9277
Record Dates: First submitted 2012-05-06; First posted 2012-05-08 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Schizophrenia
Keywords: Melatonin; Olanzapine; Metabolic side effects; Psychosis; Hyperlipidemia; Hyperglycemia; Weight gain; Diabetes
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hyperlipidemias; Hyperglycemia; Weight Gain; Diabetes Mellitus | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Melatonin (Experimental): Tablet melatonin 3 mg/day at 9 pm as intervention group for eight week
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo (with the same shape and taste as melatonin) at 9 pm as control group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Tablet melatonin 3 mg/day at 9 pm as intervention group
  Arms: Melatonin
Drug: Placebo — Placebo (with the same shape and taste as melatonin) at 9 pm as control group
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether melatonin can prevent metabolic side effects of olanzapine such as weight gain, elevated glucose concentrations and lipid abnormalities.

DETAILED DESCRIPTION:
Atypical antipsychotics including olanzapine are associated with significant metabolic side effects. Animal studies have suggested that melatonin might prevent some of the olanzapine-associated side effects. Melatonin is safe and is widely used as a sleep-promoting complement, and is not associated with side effects seen with other used drugs such as metformin.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 year
* First episode schizophrenia (DSM-IV-TR)
* Ability to take medicine orally
* Eligible for starting olanzapine

Exclusion Criteria:

* Married women who are at reproductive age
* History of taking olanzapine in the recent 3 months
* History of allergy or intolerance to olanzapine
* History of significant head trauma ( causing loss of consciousness more than 5 minutes or neurological or cognitive sequels)
* Liver, kidney, cerebrovascular or cardiovascular disease
* Diabetes, metabolic syndrome
* Cancer
* Using antiepileptic (other than benzodiazepines for sleep) , antihypertensive, anticoagulant, anti-platelet drugs
* Using inhibitors or stimulants of hepatic isoenzymes that metabolize melatonin or olanzapine (e.g. omeprazole. rifampin, fluvoxamine, ciprofloxacin, carbamazepine, modafinil)
* Delirium
* Need for administration of other antipsychotics
* Substance abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weight at week eight | Baseline and week eight

SECONDARY OUTCOMES:
Change from baseline in Triglyceride at week 4 | Baseline and week 4
Change from baseline in HDL at week 4 | Baseline and week 4
Change from baseline in LDL at week 4 | Baseline and week 4
Change from baseline in Total Cholesterol at week 4 | Baseline and Week 4
Change from baseline in weight at week 4 | Baseline and week 4
Change from baseline in Fasting blood sugar at week 4 | Baseline and week 4
Change from baseline in blood pressure at week 4 | Baseline and week 4
Change from baseline in body mass index (BMI) at week 4 | Baseline and week 4
Change from baseline in waist to hip ratio at week 4 | Baseline and week 4
Change from baseline in Positive and negative syndrome scale (PANSS) at week 4 | Baseline and week 4
Change from baseline in Positive and negative syndrome scale (PANSS) at week 8 | Baseline and week 8
Change from baseline in Triglyceride at week 48 | Baseline and week 8
Change from baseline in HDL at week 8 | Baseline and week 8
Change from baseline in LDL at week 8 | Baseline and week 8
Change from baseline in Total Cholesterol at week 8 | Baseline and Week 8
Change from baseline in Fasting blood sugar at week 8 | Baseline and week 8
Change from baseline in blood pressure at week 8 | Baseline and week 8
Change from baseline in body mass index (BMI) at week 8 | Baseline and week 8
Change from baseline in waist to hip ratio at week 8 | Baseline and week 8
Change from baseline in Insulin at week 8 | Baseline and week 8
Number of adverse events at the end of the study in each group | Baseline, week 4, and 8
Changes from baseline in HOMA-IR values at week 8 | Baseline and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jafar Modabbernia, MD, Study Chair — Guilan University of Medical Sciences
Locations (1):
- Shafa Psychiatric Hospital, Rasht, Gilan Province, Iran

REFERENCES:
- [Background] Raskind MA, Burke BL, Crites NJ, Tapp AM, Rasmussen DD. Olanzapine-induced weight gain and increased visceral adiposity is blocked by melatonin replacement therapy in rats. Neuropsychopharmacology. 2007 Feb;32(2):284-8. doi: 10.1038/sj.npp.1301093. Epub 2006 May 10. PMID 16710316
- [Background] Borba CP, Fan X, Copeland PM, Paiva A, Freudenreich O, Henderson DC. Placebo-controlled pilot study of ramelteon for adiposity and lipids in patients with schizophrenia. J Clin Psychopharmacol. 2011 Oct;31(5):653-8. doi: 10.1097/JCP.0b013e31822bb573. PMID 21869685
- [Background] Anderson G, Maes M. Melatonin: an overlooked factor in schizophrenia and in the inhibition of anti-psychotic side effects. Metab Brain Dis. 2012 Jun;27(2):113-9. doi: 10.1007/s11011-012-9307-9. Epub 2012 Apr 25. PMID 22527998
- [Derived] Modabbernia A, Heidari P, Soleimani R, Sobhani A, Roshan ZA, Taslimi S, Ashrafi M, Modabbernia MJ. Melatonin for prevention of metabolic side-effects of olanzapine in patients with first-episode schizophrenia: randomized double-blind placebo-controlled study. J Psychiatr Res. 2014 Jun;53:133-40. doi: 10.1016/j.jpsychires.2014.02.013. Epub 2014 Feb 24. PMID 24607293